CLINICAL TRIAL: NCT03505515
Title: Treatment Patterns, Clinical Outcomes, and Healthcare Resource Utilization Associated With Chinese Patients With Advanced/Metastatic Lung Cancer: a Retrospective Observational Study
Brief Title: Treatment Patterns, Clinical Outcomes, and Healthcare Resource Utilization Associated With Chinese Patients With Advanced Lung Cancer
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-693
Record Dates: First submitted 2018-04-06; First posted 2018-04-23 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer NSCLC; Small Cell Lung Cancer SCLC
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Cancer Patricipants in China: Participants with advanced/metastatic lung cancer (advanced NSCLC (IIIB/IV) and extensive disease SCLC) in China

SUMMARY:
The purpose of the study is to document real-world pattern of care, outcomes and health resource use for participants diagnosed with and receiving treatment for advanced Non-small cell lung cancer (NSCLC) and extensive disease Small cell lung cancer (SCLC) in China.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced NSCLC (IIIB/IV) and extensive disease SCLC with pathology/cytology record between 1-Dec-2013 and 30-Nov-2014
* Received inpatient treatment more than twice (inclusive) at a selected site. For hospitals with outpatient records, patients receiving oral TKI therapy and routinely (more than twice a year) followed up outpatient will be included although no inpatient records. For hospitals with outpatient chemotherapy center, patients will be include if they were prescribed with chemotherapy and routinely (more than twice a year, inclusive) followed up outpatient in the hospital
* 18 years of age or older at initial diagnosis of IIIB/IV NSCLC and extensive disease SCLC

Exclusion Criteria:

* Patients who have participated in or are attending clinical trials receiving active LC therapy
* Unknown initial diagnosis time and initial treatment time.
* For hospitals without outpatient chemo therapy center, patients who were prescribed with chemo therapy but with no inpatient records will be excluded
* Patients who received inpatient therapy for one time and were not routinely (more than twice a year, inclusive) followed up outpatient will be excluded

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with and receiving treatment for advanced NSCLC and extensive disease SCLC in China.
Sampling Method: Non-Probability Sample
Enrollment: 6205 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Proportion of participants receiving first-line systemic therapy | Approximately 36 months
  Proportion of patients receiving first-line systemic anti-cancer treatment (chemotherapy, biologic/targeted therapy)
Proportion of participants receiving second-line systemic therapy | Approximately 36 months
  Proportion of patients receiving second-line systemic anti-cancer treatment (chemotherapy, biologic/targeted therapy)
Proportion of participants receiving third-line systemic therapy | Approximately 36 months
  Proportion of patients receiving third-line systemic anti-cancer treatment (chemotherapy, biologic/targeted therapy)
Proportion of participants receiving fourth-line systemic therapy | Approximately 36 months
  Proportion of patients receiving fourth-line systemic anti-cancer treatment (chemotherapy, biologic/targeted therapy)
Distribution of first-line regimens | Approximately 36 months
  All chemotherapy, radiation and/or biologic drugs given to a patient during the first 28 days after initiation of treatment
Distribution of subsequent regimens | Approximately 36 months
  All chemotherapy, radiation and/or biologic drugs given to a patient following first-line regimen
Distribution of first-line treatment duration | Approximately 36 months
  Calculated by the difference between the treatment start date of the first observed drug in the regimen and the last observed date of the regimen
Distribution of subsequent treatment duration | Approximately 36 months
  Calculated by the difference between the treatment start date of the first observed drug in the regimen and the last observed date of the regimen
Distribution of first-line therapy completion rate | Approximately 36 months
  Completion of more than 4 cycles
Distribution of subsequent therapy completion rate | Approximately 36 months
  Completion of more than 4 cycles

SECONDARY OUTCOMES:
Distribution of patient demographic data | At baseline
Distribution of disease characteristic data | At baseline
Distribution of Overall Survival from first observed diagnosis to death | At baseline
Distribution of Overall Survival from the initiation of first-line systemic anti-cancer therapy to death | At baseline
Distribution of Overall Survival from the initiation of second-line systemic anti-cancer therapy to death | At baseline
Distribution of Overall Survival from the initiation of third-line systemic anti-cancer therapy to death | At baseline
Distribution of Overall Survival from the initiation of fourth-line systemic anti-cancer therapy to death | At baseline
Distribution of other cancer-directed therapies | Approximately 36 months
  Distribution of other cancer-directed therapies including surgery and radiation as well as supportive care
Distribution of Interval of Therapy | Up to 36 months
Distribution of Lung Cancer related direct health care costs | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Shanghai, SHG, China

REFERENCES:
- [Derived] Qiu B, Li G, Luo F, Cai X, Wu L, Chen J, Hu Y, Tang Z, Yang S, He J. Treatment patterns, clinical outcomes, and healthcare resource use associated with advanced/metastatic lung cancer in China: protocol for a retrospective observational study. Transl Lung Cancer Res. 2020 Dec;9(6):2460-2468. doi: 10.21037/tlcr-20-1269. PMID 33489806
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm